CLINICAL TRIAL: NCT05091905
Title: Patient-Titrated Automated Intermittent Boluses of Local Anesthetic vs. a Continuous Infusion Via a Perineural Catheter for Postoperative Analgesia
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Brian M. Ilfeld, MD, MS, Professor of Anesthesiology, In Residence, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Patient-Titrated Boluses cPNB
Record Dates: First submitted 2021-10-11; First posted 2021-10-25 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Pain, Acute Postoperative; Trauma Injury
MeSH Terms: conditions — Pain, Postoperative; Accidental Injuries

STUDY DESIGN:
Intervention Model Description: Randomized, Unmasked, Active-Controlled Human Subjects Clinical Trial
Masking Description: It will be impossible to mask investigators as they program the infusion pumps based on treatment group assignment; it will be impossible to mask participants as they will either be told how to titrate the bolus doses or not; and it will be impossible to mask the outcome assessor as we need to query patients on their daily bolus dose volume to track changes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Continuous Infusion (Active Comparator): Patients will receive a continuous infusion of Ropivacaine 0.2% (6 mL/hr popliteal-sciatic and 8 mL/hr infraclavicular, 4 mL patient controlled bolus with 30-minute lockout).
  Interventions: Drug: Continuous Infusion of ropivacaine 0.2%
- Titratable Automated Boluses (Experimental): Patients will receive patient-titratable intermittent boluses of Ropivacaine 0.2% (8 mL popliteal-sciatic or 11 mL infraclavicular automated bolus every 120 minutes, 4 mL patient controlled bolus with 30-minute lockout).
  Interventions: Drug: Titratable Automated Intermittent Boluses of ropivacaine 0.2%

INTERVENTIONS:
Drug: Continuous Infusion of ropivacaine 0.2% — Patients will receive a continuous infusion of Ropivacaine 0.2% (6 mL/hr popliteal-sciatic and 8 mL/hr infraclavicular, 4 mL patient controlled bolus with 30-minute lockout) will be initiated in the recovery room.
  Other Names: Perineural local anesthetic infusion
  Arms: Continuous Infusion
Drug: Titratable Automated Intermittent Boluses of ropivacaine 0.2% — Patients will receive patient-titratable intermittent boluses of Ropivacaine 0.2% (8 mL popliteal-sciatic or 11 mL infraclavicular automated bolus every 120 minutes, 4 mL patient controlled bolus with 30-minute lockout). In addition, the infusion pump will be set in a "pause" mode that delays initiation of the automated bolus doses by 5 hours (this can be over-ridden by patients if they would like to initiate their perineural infusion earlier than 5 hours). Lastly, subjects will be able to titrate the volume of their automated bolus up or down within the range of 1-16 mL.
  Other Names: Perineural local anesthetic administration
  Arms: Titratable Automated Boluses

SUMMARY:
This will be a randomized comparison of continuous local anesthetic infusion with patient controlled boluses (PCA) to patient-titratable automated boluses with patient controlled boluses (PCA) for both infraclavicular and popliteal-sciatic perineural catheters. The overall goal is to determine the relationship between method of local anesthetic administration (continuous with PCA vs. titratable intermittent dosing with PCA) for these two perineural catheter locations and the resulting pain control. The investigators hypothesize that, compared with a traditional fixed, continuous basal infusion initiated prior to discharge, perineural local anesthetic administered with titratable automated boluses at a lower dose and a 5-hour delay following discharge will (1) provide at least noninferior analgesia during the period that both techniques are functioning; and, (2) will result in a longer overall duration of administration [dual primary end points].

DETAILED DESCRIPTION:
Specific Aim: to determine the relationship between method of local anesthetic administration (continuous with PCA vs. titratable intermittent dosing with PCA) for popliteal-sciatic and infraclavicular perineural catheters and the resulting pain control.

Hypothesis: The investigators hypothesize that, compared with a traditional fixed, continuous basal infusion initiated prior to discharge, perineural local anesthetic administered with titratable automated boluses at a lower dose and a 5-hour delay following discharge will (1) provide at least noninferior analgesia during the period that both techniques are functioning; and, (2) will result in a longer overall duration of administration [dual primary end points].

This will be a randomized, controlled investigation.

Enrollment: Consenting adults undergoing painful foot and/or ankle surgery with a planned popliteal-sciatic perineural catheter insertion will be offered enrollment.

Block placement: The nerve block site will be cleaned with chlorhexidine gluconate and isopropyl alcohol (ChloraPrep One-Step, Medi-Flex Hospital Products, Inc., Overland Park, KS, USA), and a clear, sterile, fenestrated drape applied. The ultrasound probe will be readied for use and placed to visualize the short-axis (cross-section) of the target nerve. A skin wheal will be raised at the catheter-placement needle's anticipated point of entry. An 8.9 cm, 17-gauge, insulated needle (FlexTip, Arrow International, Reading, PA, USA) will be used to place all perineural catheters. The catheter-placement 17G needle will be inserted through the skin wheal, advanced in-plane beneath the US transducer and directed toward the target nerve. Normal saline (1-2 mL) will be administered via the needle to open the space around the nerve.

A flexible non-stimulating perineural catheter (FlexTip, Arrow International, Reading, PA, USA) will be inserted 2-3 cm past the needle tip. After catheter insertion, Ropivacaine 0.5% (20 mL) will be administered via the catheter under ultrasound visualization. Sensation in the treated nerve distributions will be checked for anesthetic effect up to 30 minutes following initial local anesthetic bolus. A "successful" regional block will be defined as sensory- and motor-block onset in all expected nerve distributions within the 30 minutes following the local anesthetic injection.

A saphenous nerve block with ropivacaine 0.5% (with epinephrine) may or may not be provided, depending on the surgical procedure, per standard of care.

Intraoperative: The initial local anesthetic bolus may provide complete surgical anesthesia for the procedure. Patients who desire a general anesthetic or experience a partial block that is not adequate for surgical anesthesia will receive a general anesthetic, per standard of care.

Randomization: Subjects will be randomized to one of two treatment groups: (1) titratable automated intermittent bolus or (2) continuous infusion in a computer generated 1:1 ratio using opaque envelopes opened only after successful catheter insertion is documented within 30 minutes of the local anesthetic injection.

Postoperative Procedures: Following completion of the procedure in the operating room, an infusion pump (Infutronix, Natick, Massachusetts) with a 500 mL ropivacaine 0.2% reservoir will be attached to the perineural catheter. For patients in the continuous infusion group, the pump will provide an 8 (infraclavicular) or 6 (sciatic) mL/h basal infusion and a 4 mL patient-controlled bolus with a 30-minute lockout (standard at UCSD). For patients in the titratable automated intermittent bolus group, the pump will provide an automatic 11 (infraclavicular) or 8 (sciatic) mL bolus once every 2 hours and have a 4 mL patient-controlled bolus with a 30 minute lockout. In addition, for those in the titratable automated intermittent bolus group, the infusion pump will be set in a "pause" mode that delays initiation of the automated bolus doses by 5 hours (this can be over-ridden by patients if they would like to initiate their perineural infusion earlier than 5 hours). Lastly, subjects in the titratable automated intermittent bolus group will be able to titrate the volume of their automated bolus up or down within the range of 1-16 mL.

Per standard of care, the pump will not administer more than 20 mL during each hour (below the current institutional maximum). Prior to discharge, the functioning of the infusion pump will be explained, so that they understand that they should push the bolus button if they have pain. This is accurate regardless of which treatment group the patient is randomized to, ensuring that all subjects will receive adequate analgesia.

Data Collection: Subjects will be contacted via phone for the 9 days following surgery to collect outcome measures. When 500 mL has been infused or on postoperative Day 8-whichever comes first-subjects will remove the catheter and place the pump in a pre-addressed and -stamped package for return.

Data Acquisition. Data will be gathered from the patients' electronic medical record, by telephone follow-up, and from the memory of each infusion pump. Subjects will be contacted by phone for the 9 days following surgery. Data will be recorded on paper Case Report Forms, including: patient name, medical record number, age, sex, height, weight, surgical procedure, data of procedure, anesthesiology attending overseeing/placing catheter, randomization number, whether a femoral/saphenous block was placed, if the catheter was placed per protocol, if the block set up successfully, intraoperative fentanyl, morphine and dilaudid, and the time of infusion initiation.

Statistics: The infraclavicular and popliteal-sciatic groups will be analyzed separately as two distinct analyses, each a completely separate investigation from the other. This study will be powered for two primary end points: (1) the average pain level measured with the Numeric Rating Scale queried on postoperative day 1; and (2) the duration of treatment from when the infusion pump was initially turned on until the local anesthetic reservoir was exhausted [recorded by the infusion pump memory]. The dual hypotheses will be tested with a serial testing strategy, such that Hypothesis 2 will not be formally tested unless the conclusion of Hypothesis 1 is at least "noninferiority". Following the approach described in Althunian et al, noninferiority will be assessed by comparing the lower limit of the 95% confidence interval for the difference (CB minus AB) on the NRS (range: 0 to 10) to a pre-specified noninferiority margin of 1.7 NRS units. This will provide evidence that the analgesia provided by the novel automated boluses is no worse than 1.7 NRS units compared to CB.

Baseline characteristics of the randomized groups will be summarized with means, standard deviations, and quartiles. Balance between groups will be assessed following the approach described by Schober, et al. Specifically, standardized differences will be calculated using Cohen's d whereby the difference in means or proportions is divided by the pooled standard deviation estimates. Any key variables (age, sex, height, weight, and BMI) with an absolute standardized difference >0.47 (based on Austin, 2009 with 1.96×√(2/n)=0.47) will be noted and included in a linear regression model to obtain an estimate of the treatment group differences adjusted for the imbalanced covariate(s). If residuals from the linear regression indicate violations of key assumptions (i.e. homoscedasticity or Guassian distribution), data transformations and/or alternative generalized linear models will be applied as appropriate.

Secondary outcomes will also be analyzed by Wilcoxon-Mann-Whitney test, or linear models (or generalized linear models) as appropriate with covariates for any imbalanced covariates. No multiplicity adjustments will be applied for these analyses. End points will be analyzed for each day (e.g., opioid consumption on Day 2) as well as all days combined (e.g., cumulative opioid consumption Days 1-9).

Sample size estimate: Power is simulated based on the distribution of pain measured with the Numeric Rating Scale (NRS) observed in the "Above bifurcation" group in Monahan, et al, for the sciatic catheter group. For the infraclavicular group, we simulated NRS scores from the basal/bolus treatment from Ilfeld et al. (2004). Specifically, the investigators simulate NRS scores from a discrete distribution as depicted in Figure 2 of the IRB-approved protocol (figures unavailable in this registry). This results in an expected interquartile range of approximately 1 to 4, and a median of approximately 3 NRS units. The investigators simulated 1,000 trials in which the two groups, n=35 per group, were assumed to follow the same discrete distribution, submitted each trial to a Wilcoxon-Mann-Whitney test, and derived 95% confidence intervals (Bauer 1972; Hothorn, et al. 2008). Out of the 1,000 trials, 792 (79.2%) correctly resulted in a conclusion of non-inferiority; suggesting that the probability that the trial correctly concludes non-inferiority is about 80% when the groups follow exactly equivalent distributions.

If the test for Hypothesis 1 concludes noninferiority, the investigators will test for a difference in overall duration of administration again using the Wilcoxon-Mann-Whitney test. Power is approximated by a two-sample t-test calculation. Assuming a standard deviation of SD=37 hours (corresponding to an interquartile range of 50 to 100 hours), the investigators expect that a sample size of n=35 provides 80% power to detect a mean group difference of 25 hours with a two-sided alpha of 5%.

Total enrollment: For each of the popliteal-sciatic and infraclavicular catheters, 70 subjects plus 30 for misplaced catheters or subjects otherwise unable to be randomized; and subjects who withdraw. This allows for a possible total of 100 subjects in each sub-study, and therefore a combined total of a maximum of 200 enrolled patients.

ELIGIBILITY:
Inclusion Criteria:

- patients undergoing ulnar and/or radial fracture open reduction internal fixation or painful foot and/or ankle surgery with a planned infraclavicular or popliteal sciatic perineural catheter, respectively, for postoperative analgesia

Exclusion Criteria:

* daily opioid use within the previous 4 weeks
* clinical neuro-muscular deficit of either the brachial plexus (infraclavicular) or sciatic nerve (sciatic catheters) and its branches and/or innervating muscles
* morbid obesity [body mass index > 35 kg/m2]
* surgery outside of the ipsilateral sciatic and saphenous nerve distributions for sciatic catheters [e.g., iliac crest bone graft]
* pregnancy
* incarceration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2022-02-14 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Average Pain queried on First postoperative day | Postoperative day 1
  Rated 0-10 on numeric rating scale the average pain from the recovery room until the data collection call (0=no pain, 10=worst imaginable pain)
Duration of local anesthetic administration | The first 8 days postoperatively
  The duration of treatment from when the infusion pump was initially turned on until the local anesthetic reservoir was exhausted [recorded by the infusion pump memory]

SECONDARY OUTCOMES:
Worst pain | Each of 9 days postoperatively
  Rated 0-10 on numeric rating scale over the previous 24 hours (0=no pain, 10=worst imaginable pain)
Average pain | Each of 9 days postoperatively
  Rated 0-10 on numeric rating scale over the previous 24 hours (0=no pain, 10=worst imaginable pain)
Least pain | Each of 9 days postoperatively
  Rated 0-10 on numeric rating scale over the previous 24 hours (0=no pain, 10=worst imaginable pain)
Current pain | Each of 9 days postoperatively
  Rated 0-10 on numeric rating scale (0=no pain, 10=worst imaginable pain)
Opioid consumption | Each of 9 days postoperatively
  Opioid consumption during the 24 h period prior to the data collection phone call
Cumulative opioid consumption | The first 9 postoperative days following recovery room discharge
  Cumulative opioids consumed during the first 9 postoperative days
Awakenings due to pain | The first 9 postoperative evenings queried on the following day
  The number of awakenings from sleep due to pain the previous night
Satisfaction with analgesia | The first 9 postoperative days
  0-10 scale with 0=very dissatisfied and 10=completely satisfied for the previous 24 hours
Numbness in foot and ankle for popliteal-sciatic catheters (or hand/forearm for infraclavicular catheters) | Each of 9 postoperative days
  Rate 0 = normal to 10 = insensate for the previous 24 hours
Pain Interference Subscale of the Brief Pain Inventory | Each of 9 days postoperatively
  Interference with physical and emotional functioning using a 0 to 10 scale (where 0 indicates no interference and 10 indicates complete interference). The seven interference questions involve general activity, mood, walking ability, normal work activities (both inside and outside of the home), relationships, sleep, and enjoyment of life. These seven functioning questions are combined to produce an interference subscale (0 to 70).

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, MD, MS, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No